CLINICAL TRIAL: NCT06675331
Title: Medically Utilized Tailored Traditional Meals to Optimize Nutrition in Heart Failure Pilot Trial
Brief Title: Mutton Heart Failure Food is Medicine Pilot
Acronym: Mutton-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Indian Health Service (IHS) (U.S. Federal Agency); Brigham and Women's Hospital (Other); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10072024
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: indigenous; food is medicine; Traditional Foods; Nutrition Security; Navajo
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal delivery program (Experimental): Patients will receive 2 meals daily (14 meals weekly) of medically-tailored meals incorporating traditional Navajo foods, followed by a cooking class at the end of the meal program (meals provided for 4 weeks)
  Interventions: Other: Medically Tailored Meal Program with Traditional Navajo Foods

INTERVENTIONS:
Other: Medically Tailored Meal Program with Traditional Navajo Foods — Patients will receive medically-tailored meals incorporating local traditional Navajo foods

SUMMARY:
Study subjects with heart failure will receive either pre-prepared, home-delivered DASH/SRD-compliant meals incorporating local Navajo traditional foods or usual care for 30 days (14 meals weekly).

DETAILED DESCRIPTION:
The American Indian and Alaska Native population has experienced significant cardiovascular health disparities compared with other racial and ethnic groups in the U.S. [1] Heart failure, in particular, causes significant morbidity and mortality in Navajo Nation. For many Navajo patients, similar to other American Indian populations, food insecurity is a major driver of health disparities. [2][3] In fact, qualitative data from our heart failure patient advisory committee have found that 89% of patients with heart failure believe nutrition insecurity is a major barrier to optimal health. Dietary factors are believed to be an important cause of hospitalizations in patients with heart failure and cardiovascular outcomes. There is increasing evidence that direct dietary support, such as produce prescription or provision of medically tailored meals may improve cardiovascular outcomes and disease-specific quality of life. Furthermore, there has been an increased focus in Indigenous communities to reclaim traditional indigenous foods to improve health. However, more evidence of the benefit of traditional Indigenous foods for cardiovascular health is needed.

We, therefore, in discussion with community members and tribal partners at two Indian Health Service (IHS) sites in Navajo Nation, will implement and evaluate the effectiveness of a medically and Native-sourced culturally tailored meal delivery program to improve outcomes in heart failure in rural Navajo Nation. This study will include two phases, with a phase I pilot feasibility study, followed by phase II-a comparativeness effectiveness randomized controlled trial to compare the implementation of our medically and culturally tailored meal delivery program compared to usual care. For phase I, we will conduct a one-arm pilot trial of the MUTTON-HF intervention to determine 1) feasibility of the intervention and outcome assessment and 2) acceptability of the intervention and 3) fidelity of the intervention. We will enroll 20 patients to receive medically tailored meals (14 meals weekly) for 30 days to inform the phase II comparativeness effectiveness trial.

Phase I outcomes will include implementation outcomes such as feasibility and acceptability of the intervention including the various delivery mechanisms and meals as measured by quantitative (i.e. % meals delivered and % meals received by patient) and qualitative methods, of outcome assessment including surveys and laboratory evaluation (% with completed outcome assessment), and fidelity of intervention as measured by quantitative (% meals consumed). We will additionally measure feasibility and acceptability of supporting local food systems by measuring % meals with locally sourced produce and meat, and % sourced from Navajo farmers and ranchers specifically. We will also explore implementation outcomes with community partners including farmers, growers, ranchers, food pantry.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* ICD I50* diagnosis
* Clinical encounter in last 12 months
* Primary care physician at the two IHS sites
* Hospitalization (any-cause) within last 12 months

Exclusion Criteria:

* Hospice care
* Living in acute rehabilitation or skilled nursing facility
* Living outside the Gallup Service Unit (outside 50-mile catchment area)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Feasibility: Percentage of meals successfully received by the patient | 30 days
  Proportions of meals that were successfully picked up or received by the patient. We have determined that >70% would count as success/feasibility of the intervention.

SECONDARY OUTCOMES:
Cultural Connectedness Scale-California | Baseline, 30 Days
  The Cultural Connectedness Scale (CCS) was developed in Canada by First Nations/Indigenous persons for First Nations/Indigenous persons. The 29-item CCS consists of three sub-scales: identity, traditions, and spirituality. This scale ranges from 0-40, with 40 indicating higher levels of cultural connectiveness.
Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | Baseline, 30 Days
  This is a validated score for evaluating quality of life and symptom measures in heart failure patients. Score ranges from 0-100, with 0 meaning very poor quality of life/symptoms and health status, 100 meaning excellent quality of life/symptom burden/health status.
USDA Adult Food Security: Six Item short Form survey | Baseline, 30 Days
  The six-item short form of the survey module and the associated Six-Item Food Security Scale were developed by researchers at the National Center for Health Statistics in collaboration with Abt Associates Inc.
Hospitalization or Emergency Department Visit | 90 Days
  Hospitalization or Visit to Emergency Department (All-cause)
Laboratory Biomarker Data | Baseline, 30 Days
  Albumin, prealbumin, creatinine, NT-proBNP, HbA1c, Total cholesterol, LDL-C, HDL-C, Triglycerides, CRP
Weight/Body Mass Index | Baseline, 30 Days
  weight and BMI
Emergency Room Visits | 90 Days
  ER visits: All cause
ER visits or hospitalizations | 180 days
  All cause
ER visit for Heart Failure | 90 Days
  ER visit for volume overload or HF symptoms
Heart Failure Hospitalizations | 90 days
  Hospitalizations for heart failure specifically
Feasibility: Percentage of meals delivered successfully to the Gallup Food Pantry | 30 days
  Proportions of meals that were successfully delivered to the Gallup Food Pantry by our community partner and Native-run Kitchen
Feasibility of Intervention: Delivery/Pick-Up | 30 days
  We will survey patients post-intervention with question to assess feasibility: "I would rate getting the meals (either picking up or delivery): Very easy, Somewhat easy, Neither easy nor difficult, Somewhat difficult, Very difficult.
Acceptability of the Intervention (AIM) Measure | 30 days
  We will evaluate acceptability of the intervention among the patients through quantitative assessment using the validated acceptability of the intervention (AIM) measure
Net Promoter Score | 30 days
  We will also assess acceptability of the intervention through assess the Net Promoter Score (i.e. how likely is it that you would recommend this program to a community member?"), which is a scale 1 (highly unlikely) to 10 (highly likely).
Fidelity: Consumption | 30 days
  Patients will also rate meals from 1-5 and the amount of the meal they consumed (none [or only a few bites], less than half, about half, most, or all)
Acceptability: Taste | 30 days
  Patients will also be surveyed post-intervention the following questions to assess acceptability: How would you rate the meals overall, in terms of taste (excellent, good, average, below average, bad?"
Qualitative measures of feasibility and acceptability | 30 days
  We will also perform semi-structured interviews of patients to assess feasibility and acceptability through qualitative methods. Semi-structured interviews will be guided by the Consolidated Framework for Implementation Research (CFIR), and we will explore multiple constructs within each CFIR domain that are hypothesized by the study team and based on existing literature to be relevant to acceptability and feasibility of the program
Feasibility of Supporting Local Food Systems | 30 days
  We will assess feasibility among our community partners by assessing the validated feasibility of the intervention measure (FIM) among our food pantry partners.
Feasibility: Local Food Sourcing | 30 days
  We will also assess the % of meals that include locally sourced ingredients, % of meals sourced by Native suppliers/farmers (produce), % of meals soured by Native ranchers (meat)
Feasibility of Outcome Assessment | 30 days
  We will determine the proportion of patients that completes baseline, as well as post-implementation survey and laboratory data.
  We will consider ≥ 80% completion rates as a success.
Fidelity of Intervention | 30 days
  We will assess fidelity of the intervention by evaluating:
  * We will have patients' complete food diaries for 3 days during week 1 and week 4 of the intervention.
  * % of meals consumed: Patients will also fill out meal cards weekly with percent consumed (None [or a few bites], ¼, ½, ¾, all [or nearly all]).
    § We will stratify meals consumed by whether the meal used traditional Diné ingredients or not.
  * We will additionally survey participants post-intervention the following:
    * In terms of leftovers, how much of the meals were not eaten and had to be thrown out? (all, most, about half, less than half, none).
      * We will consider ≥ 70% meals consumed (at least ½ or more of the meal) or ≥70% indicating they ate "most" or more of the meals as a success
Adoption of Intervention | 30 days
  We will survey participants post-intervention the following using a Likert scale:
  * How likely is it that this program will change your diet to be healthier moving forward? (very likely, somewhat likely, neither likely nor unlikely, somewhat unlikely, very unlikely)
  * How likely is it that you will add any of the meals or recipes from this program to your on-going diet in the future? (very likely, somewhat likely, neither likely nor unlikely, somewhat unlikely, very unlikely)
Diet Quality | Baseline and 30 days
  We will assess diet quality using the 10-item DSQ [10] with an addition question to assess traditional Dine food intake (During the past month, how often did you eat traditional Diné foods (such as blue corn mush, steamed, roasted or dried corn, sumac berries, mutton, local varieties of squash or beans) at baseline and at the end of the intervention.
Physical Activity | Baseline and 30 days
  We will evaluate how much physical activity/exercise patients are participating in weekly at baseline, and at 30 days by asking patients to estimate the number of minutes weekly that they are participating in formal exercise or physical activity.
General Health Status | Baseline and 30 days
  We will evaluate patients' general health status using a single general health status question (would you say that in general your health is excellent, very good, good, fair, or poor) at baseline and post-intervention
KCCW12-PL Physical Limitation Score | 30 days
  Subsection of KCCQ-12 Summary
KCCQ12-PL Physical Limitation Score | 30 days
  Subsection of KCCQ12 looking at physical limitation
KCCQ12-SF Symptom Frequency Score | 30 Days
  Subsection of KCCQ-12 looking at frequency of symptoms
KCCQ-QL | 30 Days
  Subsection of KCCQ-12 that looks at quality of life
KCCQ-SL Social Limitation Score | 30 days
  Subsection of KCCQ-12 looking at social limitation

OTHER OUTCOMES:
Medication and Medical Therapy Adherence | 30 days
  Additional exploratory outcomes will prescription rates for all medication as well as guideline-directed medical therapy specifically (for heart failure with reduced ejection fraction this would include ACEi/ARB/ARNI, Beta-blocker, SGLT2 inhibitors, and mineralocorticoid receptor antagonist; for HFpEF this would include SGLT2 inhibitors).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Eberly, MD, MPH, Principal Investigator — Indian Health Service (IHS)
Locations (1):
- Tohatchi Health Clinic, Tohatchi, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
Data is tribally owned data and is protected under Navajo Nation Human Research Review Board regulations.

REFERENCES:
- [Derived] Eberly LA, George C, Sandman S, Bex D, Chandra M, Shultz K, Tennison A, Wickre R, Wickre B, Morgan L, Gray L, Bolas M, Feliciano B, Damon-Mallette D, Lindsey E, Manche J, Detsoi-Smiley P, Mora P, Merino M, Shin SS. Feasibility of an Indigenous Food Is Medicine Program for Patients With Heart Failure in Rural Navajo Nation: The MUTTON-HF Nonrandomized Clinical Trial. JAMA Netw Open. 2026 Feb 2;9(2):e2556117. doi: 10.1001/jamanetworkopen.2025.56117. PMID 41649816
- See also: Trial website — http://www.muttonhf.com